CLINICAL TRIAL: NCT00004029
Title: A PHASE I TRIAL OF RECOMBINANT VACCINIA VIRUS THAT EXPRESSES PSA IN PATIENTS WITH ADENOCARCINOMA OF THE PROSTATE
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065275; DFCI-96079; NCI-T95-0086H
Record Dates: First submitted 1999-12-10; First posted 2004-08-30 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2006-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim

ARMS (1):
- Arm I (Experimental): atients in cohorts of 3-6 receive 3 vaccinations with rV-PSA at 4-week intervals (days 1, 29, 57, and 85) in the absence of disease progression or unacceptable toxicity. Response assessment is performed at eight weeks. Patients who discontinue therapy prior to eight weeks are considered unevaluable for response. If dose limiting toxicity is observed in 2 of 6 patients entered at a dose level, no further patients are entered at that level and the MTD is defined as the preceding dose level. Ten additional patients are treated at the MTD and receive granulocyte-macrophage colony-stimulating factor (GM-CSF) administered subcutaneously on day -1 through day 2 of each cycle. Patients who are HLA-A2 positive, have received all 3 rV-PSA vaccinations without unacceptable toxicity, and have been off study for at least 30 days due to disease progression may continue treatment with rV-PSA at the highest dose level and the addition of GM-CSF.
  Interventions: Biological: recombinant viral vaccine therapy; Biological: sargramostim

INTERVENTIONS:
Biological: recombinant viral vaccine therapy
Biological: sargramostim

SUMMARY:
Phase I trial to study the effectiveness of vaccine therapy in treating patients with metastatic prostate cancer. Vaccines may make the body build an immune response to kill tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Assess the toxicity associated with repeated vaccination with recombinant vaccinia virus expressing prostate-specific antigen (rV-PSA) in patients with metastatic adenocarcinoma of the prostate.

II. Determine the optimal dose of rV-PSA given at monthly intervals based on cellular and hormonal immunity.

III. Determine whether vaccination with rV-PSA is associated with anti-tumor activity.

IV. Determine whether granulocyte-macrophage colony-stimulating factor (GM-CSF) has an effect on cellular and humoral immunity different from rV-PSA, and whether the addition of GM-CSF has enhanced antitumor effect compared to rV-PSA alone.

OUTLINE: This is an open label, dose escalation study.

Patients in cohorts of 3-6 receive 3 vaccinations with rV-PSA at 4-week intervals (days 1, 29, 57, and 85) in the absence of disease progression or unacceptable toxicity. Response assessment is performed at eight weeks. Patients who discontinue therapy prior to eight weeks are considered unevaluable for response. If dose limiting toxicity is observed in 2 of 6 patients entered at a dose level, no further patients are entered at that level and the MTD is defined as the preceding dose level. Ten additional patients are treated at the MTD and receive granulocyte-macrophage colony-stimulating factor (GM-CSF) administered subcutaneously on day -1 through day 2 of each cycle. Patients who are HLA-A2 positive, have received all 3 rV-PSA vaccinations without unacceptable toxicity, and have been off study for at least 30 days due to disease progression may continue treatment with rV-PSA at the highest dose level and the addition of GM-CSF.

Patients are followed monthly for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven adenocarcinoma of the prostate with evidence of metastatic disease based on any of the following:

  * Lymph node positive and PSA at least 10 ng/mL
  * Bone scan positive and PSA at least 10 ng/mL
  * PSA at least 2 ng/mL and rising following radical prostatectomy
  * PSA at least 10 ng/mL following radiotherapy
* No symptomatic metastatic disease (bony pain)

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0 or 1
* WBC greater than 2,000/mm3
* Platelet count greater than 100,000/mm3
* Bilirubin less than 2.0 mg/dL
* AST less than 4 times normal
* Creatinine less than 2.0 mg/dL
* Must be type HLA-A2 Prior vaccinia (smallpox) exposure required
* At least normal delayed type hypersensitivity to mumps and Candida
* At least normal CD4:CD8 ratio (greater than 1)
* At least normal lymphocyte proliferation testing (to Con A)
* At least normal immunoglobulin levels
* No evidence of altered immune responsiveness or autoimmune syndromes (e.g., scleroderma, systemic lupus erythematosus)
* No HIV antibody No prior splenectomy
* No known allergy to eggs
* No active extensive skin disorders (e.g, psoriasis, burns, impetigo, disseminated zoster)
* No other serious intercurrent illness
* No active infections unless cleared and at least 3 days since antibiotic therapy
* No close contact for 2 weeks after each vaccination with the following people:

  * Children less than 3 years old
  * Pregnant women
  * Individuals with eczema or skin conditions listed above
  * Immunosuppressed individuals

PRIOR CONCURRENT THERAPY:

* No concurrent biologic therapy
* No prior chemotherapy for metastatic disease
* No prior hormone therapy for metastatic disease
* Neoadjuvant hormone therapy prior to prostatectomy or radiotherapy allowed
* No concurrent steroids or hormonal medications
* Prior radiotherapy allowed
* Prior surgery allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1996-12; Primary Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W. Kufe, MD, Study Chair — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Eder JP Jr, Kantoff PW, Bubley GJ, et al.: A phase I trial of recombinant prostate specific antigen expressing vaccinia virus vaccine, PROSTVAC (rV-PSA) in advanced prostate cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A1692, 439, 1999.
- [Result] Eder JP Jr, Kantoff PW, Bubley GJ, et al.: A phase I trial of recombinant vaccinia virus, PROSTVAC that expresses prostate specific antigen (rV-PSA) as a vaccine in men with advanced prostate cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A1672, 434, 1998.